CLINICAL TRIAL: NCT04388332
Title: Comparison of Clinical Outcomes Following ACDF With Instrumentation Using Structural Allograft vs. Tritanium C
Brief Title: ACDF Using Structural Allograft vs. Tritanium C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Stryker Spine (Industry)
Responsible Party: Principal Investigator, Nestor Tomycz, Assistant Professor, Department of Neurosurgery, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Stryker IIT
Record Dates: First submitted 2020-04-02; First posted 2020-05-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease
Keywords: Tritanium C; Structural Bone Graft; Anterior Cervical Discectomy and Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: retrospective/prospective observational, two arm study - 40 patients in retrospective cohort (data collection from previous procedure) compared to 20 patients in Prospective cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Retrospective (Active Comparator): 40 patients that received one or two level ACDF structural allograft with plates with autograft and /or allograft comprised of cancellous and/or corticocancellous bone chips.
  Interventions: Procedure: Structural allograft
- Prospective (Experimental): 20 patients who are receiving Tritanium C as standard of care.
  Interventions: Device: Tritanium C

INTERVENTIONS:
Procedure: Structural allograft — Subjects that have received ACDF structural allograft with plates with autograft and/or allograft comprised of cancellous and/or corticocancellous bone chips
  Arms: Retrospective
Device: Tritanium C — Subjects will receive the Tritanium C anterior cervical cage which is intended to be used with autogenous or allogenic bone graft comprised of cancellous and/or corticocancellous bone graft
  Arms: Prospective

SUMMARY:
This is an observational, descriptive, prospective and retrospective data collection study. The purpose of this study is to observe radiographic outcomes of patients who will undergo anterior cervical discectomy and fusion (ACDF) utilizing Tritanium C (Stryker Spine). The rate of fusion success and adverse events will be compared retrospectively to patients who underwent instrumented ACDF utilizing structural allograft bone with plates.

DETAILED DESCRIPTION:
Retrospective Cohort: A maximum of 200 patients that received one or two level ACDF structural allograft with plates with autograft and/or allograft comprised of cancellous and/or corticocancellous bone chips at AHN in the past will retrospectively be screened for inclusion into a pool of potential candidates for the retrospective cohort. Patients will be included in this preliminary pool if the following information are available: age (at surgery), sex, body mass index (at surgery), no smoking at baseline, number of levels operated on, which specific levels were operated on, standard of care clinic follow-up at 6 and 12 months (3 month visit not required) and imaging that can be used to assess fusion at baseline, 6 and 12 months (3 month imaging not required). If available, NDI and VAS, questionnaires completed during baseline and post-op visits will be collected.

This pool of retrospective cohort candidates will be used to match the patients in the prospective cohort to patients treated with structural allograft using a 1:2 ratio. Thus, 40 patients will ultimately be included in the retrospective cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age, ≤ 80 years of age
2. Subject is skeletally mature
3. Subject is diagnosed with degenerative disc disease (DDD) at one level or two contiguous levels from the C2 -T1 disc
4. Subject has received six weeks of non-operative therapy i.e. injections, physical therapy, oral steroids
5. Subject understands the conditions of enrollment and is willing to sign and date the Informed Consent (Prospective study)
6. Subjects that will prospectively undergo one or two level anterior cervical discectomy and fusion with Tritanium C (Prospective study)
7. Subjects that underwent one or two level anterior cervical discectomy and fusion with either standard of care structural allograft bone at any AHN facility from 01/01/2016 to 08/14/2023 (Retrospective study) • Note that these patients will be followed for a maximum of one year (up to 08/14/2024 for a patient enrolled at the end of this inclusion period)

Exclusion Criteria:

Patients may not be enrolled in the study if any of the following exclusion criteria are present:

1. Presence of an infection systemic or local
2. Presence of marked local inflammation
3. Subject has any abnormality present which affects the normal process of bone remodeling including, but not limited to, severe osteoporosis involving the spine, bone absorption, osteopenia, primary or metastatic tumors involving the spine, active infection at the site or certain metabolic disorders affecting osteogenesis
4. Use of bone growth stimulator
5. Subject has prior fusion at the levels to be treated
6. Subject has any neuromuscular deficit
7. Subject has any condition of senility, mental illness, or substance abuse
8. Subject has any other medical or surgical condition which would preclude the potential benefit of spinal implant surgery in the judgement of the PI
9. Subject has rapid joint disease, bone absorption, osteopenia, osteomalacia, and/or osteoporosis. Subject is pregnant or plans to become pregnant during the course of the study.
10. BMI≥40 kg/m2
11. Subject uses chronic corticosteroids
12. Subjects with current active psychiatric diagnosis or a personality disorder likely to interfere with the study
13. Subjects who smoke and do not plan to quit
14. Mental or neuromuscular disorder which would create an unacceptable risk of fixation failure or complications in postoperative care
15. Subject has any open wounds
16. Subject has inadequate tissue coverage over the operative site
17. Subject may be sensitive to titanium materials
18. Subject is missing 6 and/or 12 month clinical or radiographic follow-up (Retrospective study)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to the presence of fusion | 3 months post-operatively
  Antero-posterior and lateral plain radiographs
Time to the presence of fusion | 6 months post-operatively
  Antero-posterior and lateral plain radiographs
Time to the presence of fusion | 12 months post-operatively
  Antero-posterior and lateral plain radiographs

SECONDARY OUTCOMES:
Neck disability | Baseline, 3, 6, and 12 months post-operatively
  Neck Disability Index (NDI): Subjects will designate a statement that best describes their level of disability for each section of the survey. Statements are then ranked from 0-5, where 0 is a better outcome and 5 is a worse outcome. All rankings are totaled for a final score.
Neck and arm pain | Baseline, 3, 6, and 12 months post-operatively
  Visual Analog Scale (VAS) for neck and arm pain: Subjects will designate a score to represent their pain from 0 to 10. 0 is indicative of no pain and 10 is indicative of the worst possible pain.
Incidence of sensory deficits | Baseline, 3, 6, and 12 months post-operatively
  Yes or no response to: Sensory deficit at the surgical level, sensory deficit at an adjacent level to the surgical level, sensory deficit at a different level to the surgical level, any sensory deficit during follow-up
Incidence of motor deficits | Baseline, 3, 6, and 12 months post-operatively
  Yes or no response to: Motor deficit at the surgical level, motor deficit at an adjacent level to the surgical level, motor deficit at a different level to the surgical level, any motor deficit
Rate of Adverse Events | Day of surgery, 3, 6 and 12 month post-operatively
  Adverse Event assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Tomycz, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- Allegheny Health Network, Pittsburgh, Pennsylvania, United States